CLINICAL TRIAL: NCT04660214
Title: Minimally Invasive Endoscopic Treatment of Zenker's Diverticulum Comparing LigaSureTM vs SB-Knife.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Mª Henar Núñez Rodriguez, MD PhD, Principal Investigator, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI208-20
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Zenker Diverticulum; Minimally Invasive Surgical Procedures; Endoscopy
MeSH Terms: conditions — Zenker Diverticulum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vessel sealing device (Active Comparator): Endoscopic diverticulectomy is performed with the LigaSure (TM) device
  Interventions: Device: septotomy
- Dissecting Knife device (Active Comparator): Endoscopic diverticulectomy is performed with the SB-Knife(TM) device
  Interventions: Device: septotomy

INTERVENTIONS:
Device: septotomy — endoscopic diverticulotomy

SUMMARY:
The main purpose of this trial is to evaluate two devices used in the treatment of Zenker Diverticulum using flexible endoscopy (LigaSure and SB-knife). Analyze the technical success, clinical success, relapses, complications, and the mean procedure time with each device prospectively in order to transfer objective and uniform results to routine clinical practice.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will be randomized on the day of the procedure using a computer system that generates a table of random numbers, to perform endoscopic diverticulotomy using a LigaSure device (LS 1500, Covidien; Medtronic, Minneapolis, MN, USA) or with Stag Beetle (SB) knife standard (Sumitomo Bakelite Co. Tokyo, Japan).

Prophylactic intravenous antibiotic therapy is administered prior to the procedure and will be performed under deep sedation with control by an endoscopist or anesthesiologist in the cases indicated.

Gastroscopy will be performed to identify Zenker's diverticulum, and isolate the septum under endoscopic control using a diverticuloscope or flexible overtube (ZD overtube, ZDO 22/30 Cook Medical), after placing a guide (0.035 ", 450 cm Jagwire, Boston Scientific, Natick MA, USA) in the esophageal lumen. The overtube has two leaflets at one of its ends, a longer one that is placed in the esophageal lumen and the short leaflet is placed in the diverticulum. In those cases in which it is not possible to place the diverticuloscope, the septum will be isolated with the help of a cap on the end of the endoscope. In these cases, the device used will always be the SB-Knife since it is not possible to use the LigaSure and they will be excluded from the study analysis.

The time of the procedure will be counted from when the overtube is placed until it is removed after diverticulotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endoscopically confirmed Zenker's diverticulum and presenting symptoms related to it.
* Those who complete the symptom and quality of life questionnaires.
* They must sign informed consent.

Exclusion Criteria:

* Previous treatment of Zenker's Diverticulum
* Those for whom Zenker's diverticulum is ruled out at endoscopy.
* Chewing disorders and/or dysphagia secondary to neurological pathology and Oesophageal motility disorders
* Those who do not want to participate in the study and/or who do not sign the informed consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the technical success of endoscopic diverticulotomy with SB-Knife and LigaSure | At the moment of the procedure
  Technical success: achieving septotomy of the mucosa and transverse muscle fibers of the diverticulum septum.
Evaluate clinical success of endoscopic diverticulotomy with SB-Knife and LigaSure | One month after the procedure
  Clinical success: disappearance of symptoms or their improvement one month after treatment, evaluated using the Eating-Assessment Tool-10 (>=3 pathological) and Dakkak and Bennett scales (0: asymthomatic; 4 aphagia)

SECONDARY OUTCOMES:
Analyze the mean procedure time with each of the two endoscopic techniques | At the end of the recruitment
  The procedure time will be counted from the overtube is placed until it is removed after diverticulectomy
Analyze immediate and delayed complications with SB-Knife and LigaSure | one month after the procedure
  Complications during the procedure and post-procedure the first 14 days after the procedure):
  * bleeding (decrease in Hb with hypotension and / or tachycardia and need for a gastroscope and hospital admission) (endoscopically controlled or if surgical treatment is required)
  * perforation: endoscopic control or surgical treatment
  * odynophagia or neck pain (VAS Scale)
  * Any complication that requires prolonging the hospital stay.
  Late complications (from the 15th day and during the first month):
  * Haemorrhage that requires endoscopic / surgical treatment or hospital admission for its control
  * Oesophageal perforation (conservative or surgical treatment): cervical emphysema, air in the mediastinum.
  * Pain that requires hospital admission
Determine the recurrence rates and the mean time to recurrence for each of the techniques | at least three months after the procedure
  Recurrence: reappearance of symptoms (dysphagia, cough ...) after their disappearance or worsening, reflected in an increase in the scores of the Dakkak and Bennett scales (score ≥1 or increase of 1 point) and EAT -10 (EAT-10 score ≥3 or 3-point increase from previous score).

CONTACTS AND LOCATIONS:
Overall Officials: Mª Henar Núñez-Rodriguez, MD PhD, Principal Investigator — Gastroenterology Department, Hospital Rio Hortega
Locations (1):
- Mª Henar Núñez Rodriguez,, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No